CLINICAL TRIAL: NCT07332065
Title: The Effect of Mandala Coloring on Menopausal Symptoms, Sexual Quality of Life, and Self-Esteem in Women During the Menopause Period
Brief Title: The Effects of Mandala Coloring on Women During Menopause
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Kevser Katkaya, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KahramanmaraşSIU-NURSİNG-KK-01
Record Dates: First submitted 2025-12-11; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Menopause; Self Esteem; Sexual Activity; Women; Menopause Symptoms
Keywords: menopause; menopause symptoms; self esteem; mandala coloring; sexual quality of life; mandala
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala coloring (Experimental): Participants will take part in 30-minute mandala painting sessions once a week for four weeks.
  Interventions: Other: Mandala coloring
- Control group (No Intervention): No intervention will be applied to participants in the control group within 4 weeks.

INTERVENTIONS:
Other: Mandala coloring — Mandala coloring is a structured creative art activity based on colouring mandala shapes, which consist of circular and symmetrical patterns, increasing focus and promoting relaxation. As one of the art therapies, mandala colouring can have a therapeutic effect on individuals.
  Other Names: Mandala art activity
  Arms: Mandala coloring

SUMMARY:
The aim of this clinical study is to determine the effect of mandala coloring on menopausal symptoms, sexual quality of life, and self-esteem in women during menopause period. The main questions the study aims to answer are as follows:

1. Does mandala coloring reduce the severity of menopausal symptoms in women?
2. Is there an increase in self-esteem levels among women who participate in mandala coloring after the intervention?
3. Is there an increase in the quality of sexual life among women who participate in mandala coloring after the intervention? Researchers will compare the intervention group (those who participated in mandala coloring) with the control group (those who did not participate in any intervention) to evaluate the effectiveness of mandala coloring.

Participants

* Participants in the intervention group will attend 30-minute mandala coloring sessions once a week for 4 weeks.
* Participants in the control group will not receive any intervention during the same period.
* Both groups will be assessed using a questionnaire at the beginning of the study and at the end of the 4th week (pre-test/post-test).

DETAILED DESCRIPTION:
Menopause is a natural, biological process that marks the end of a woman's fertile years. Every woman's menopause is unique. The experience, severity, duration, and physical and psychological effects of menopause are all unique. During this period, women must contend with both the processes of aging and the hormonal changes that occur during menopause. These changes can sometimes negatively impact an individual's life, reducing their quality of life. Menopausal symptoms can often appear one to two years before their last menstrual period and up to 15 years afterward. These symptoms, such as decreased sexual desire, decreased estrogen levels, mood disorders, illnesses associated with menstruation, decreased genital sensation, vaginal dryness, physical discomfort, and bone loss, can lead to a loss of sexual desire and alienate a person from their partner. This, in turn, leads to a decrease in self-esteem, a feeling of unease about one's own characteristics and ongoing physical and psychological changes. Consequently, individuals' anxiety levels increase, and their ability to cope with symptoms decreases. Studies have highlighted the benefits of alternative methods for coping with anxiety in women undergoing menopause. Music therapy and art therapy are examples. Studies have also demonstrated the therapeutic effects of mandala coloring, an art therapy activity. This study aims to examine the effects of mandala coloring on menopausal symptoms, quality of sexual life, and self-esteem in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40 and 65,
* Not having experienced menstruation for at least one year,
* Having a score of 15 or higher on the MSDS (meaning having experienced at least moderate menopause),
* Not having received hormone replacement therapy for menopausal symptoms,
* Not having undergone surgical menopause,
* Experiencing at least one vasomotor symptom of menopause (hot flashes, night sweats, sudden sweating attacks, palpitations, chills and shivering attacks, etc.).
* Being able to read, write, speak, and understand Turkish,
* Not having previously received mandala art therapy training or regularly practicing mandala coloring,
* Not having an allergy to mandala coloring materials,
* Not practicing spiritual practices such as yoga or meditation,
* Agreeing to participate in the study.

Exclusion Criteria:

* Having a physical symptom that may prevent mandala coloring,
* Having communication and perception problems,
* Having difficulty understanding or speaking Turkish,
* Having a psychiatric illness or taking psychiatric medication,
* Having experienced a loss in the last 6 months.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gender is suitable as the study is on menopausal symptoms.
Enrollment: 70 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Menopausal Symptoms | Time Frame: Fromenrollmenttotheend of intervention at 4 weeks.
  The primary outcome measure in this study is the severity of menopausal symptoms as assessed by the Menopause Rating Scale. This scale is an 11-item measure developed by Heineman et al. (1996) to assess the severity of menopausal symptoms. The minimum score that can be obtained on the scale is 0, while the maximum score is 44. An increase in the score obtained from the scale indicates an increase in the severity of the complaints experienced, while also showing that quality of life has been negatively affected. In this study, the validity and reliability of the scale in Turkish were conducted by Can Gürkan (2005). The Turkish version of the scale will be used. Within the scope of the current study, it is expected that women in menopause who engage in mandala coloring will show improvement in menopause symptoms. In other words, the Menopause Rating Scale scores of women in the experimental group will be lower than those of women who do not practice mandala coloring.

SECONDARY OUTCOMES:
Sexual Quality Of Life | Time Frame: From enrollment to the end of intervention at 4 weeks.
  In this study, the secondary outcome measure is the level of sexual quality of life assessed using the Sexual Quality of Life Scale. The scale, developed by Symonds et al. (2005), consists of 18 items designed to measure women's sexual quality of life. Participants are expected to respond to the items based on their sexual life over the past four weeks. The lowest possible score on the scale is 18, and the highest possible score is 108. A higher score on the scale indicates a better quality of sexual life. The Sexual Quality of Life Scale - Female Turkish Form will be used in this study. Its validity and reliability in Turkish were conducted by Gölbaşı (2010). Within the scope of the current study, it is expected that women in menopause who practice mandala coloring will show an increase in their sexual life quality. In other words, the Sexual Life Quality Scale scores of the women in the experimental group are higher than those of women who do not practice mandala coloring.
Self-Esteem | Time Frame: From enrollment to the end of intervention at 4 weeks.
  Another secondary outcome measure in this study is the level of self-esteem, assessed using the Coopersmith Self-Esteem Inventory Scale. The scale was developed by Stanley Coopersmith (1967). It consists of 25 items with opposite responses such as "Like me" or "Not like me." The content includes the person's outlook on life, family relationships, social relationships, and resilience. The lowest possible score on the scale is 0, and the highest is 25. A low score on the scale indicates low self-esteem, while a high score indicates high self-esteem. Turkish reliability and validity studies were conducted by Aksoy (1992) and Pişkin (1997). Within the scope of the study, it is expected that women in menopause who practice mandala coloring will experience an increase in their self-esteem levels. In other words, the scores obtained by the women in the experimental group on the Coopersmith Self-Esteem Inventory Scale are higher than those of women who do not practice mandala coloring.

IPD SHARING:
Plan to Share IPD: No